CLINICAL TRIAL: NCT05556213
Title: Estimation of Plasma Levels of MicroRNA 125b-5p and Transvaginal Ultrasonography May Spare Laparoscopy for Staging of Endometriosis
Brief Title: The Relation Between MiR-125b-5p and Staging of Endometriosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Hagars, Assistant professor of gynecology, Tanta University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 35617/8/22
Record Dates: First submitted 2022-09-24; First posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Active Comparator)
  Interventions: Procedure: laparoscopic examination
- Control (Active Comparator)
  Interventions: Diagnostic Test: Blood sampling

INTERVENTIONS:
Procedure: laparoscopic examination — laparoscopic examination for staging of endometriosis
  Arms: Patients
Diagnostic Test: Blood sampling — Blood sample to detect endometriosis
  Arms: Control

SUMMARY:
78 endometriosis patients presented with infertility were clinically examined and the diagnosis was assured by US imaging. The study also included 11 control fertile women free of gynecological problems as a control for lab tests. Patients and controls gave blood samples for lab investigations. All patients underwent diagnostic abdominal laparoscopy under general anesthesia for disease staging. Quantitative determination of expression levels of genes of microRNA-125b-5p and 203a was conducted using qRT-PCR.

ELIGIBILITY:
Inclusion Criteria:

* Patients who presented clinical pictures suggestive of EM disease

Exclusion Criteria:

* Patients with previous pelvic or abdominal surgery that may hinder the laparoscopic examination,
* patients who were suspicious of having malignancy elsewhere in the body region,
* pregnant women,
* patients who had diabetes mellitus,
* body mass index (BMI) of >30 kg/m2, coagulopathies, and autoimmune disorders.

Ages: 22 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Validity of Plasma expression level | two weeks
  the diagnostic validity of estimation of plasma expression levels of MiR-125b-5p and 203a for diagnosis and staging of endometriosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta university, Tanta, El-Gharbyia, Egypt